CLINICAL TRIAL: NCT04541576
Title: Prospective, Non-Randomized, Controlled, Multicenter Feasibility Study of the Merit WRAPSODY™ Endovascular Stent Graft for Treatment of Central Venous Outflow Circuit Stenosis or Occlusion in Hemodialysis Patients
Brief Title: The Merit WRAPSODY Central Feasibility Study
Acronym: WAVE Central
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA Approval
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVO-P3-20-01-F
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Venous Stenosis; Venous Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- WRAPSODY Stent Graft (Experimental): All subjects will receive treatment via WRAPSODY Stent Graft Placement.
  Interventions: Device: Merit WRAPSODY Endovascular Stent Graft

INTERVENTIONS:
Device: Merit WRAPSODY Endovascular Stent Graft — Target lesion treated with stent graft placement

SUMMARY:
The purpose of the study is to demonstrate the safety and efficacy of the Merit WRAPSODY Endovascular Stent Graft for treatment of stenosis or occlusion within the dialysis access outflow circuit in the thoracic central veins

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent
* Subject is male or female, with an age ≥ 18 years at date of enrollment.
* Subject is willing to undergo all follow-up assessments.
* Subject has a life expectancy ≥ 12 months.
* Subject is undergoing chronic hemodialysis.
* Subject has either a mature AVF or AVG in the arm.
* Target lesion(s) involves a non-stented restenotic lesion.
* Target lesion has ≥50% stenosis.
* Target lesion(s) reference vessel diameter is between 5.0 mm and 14.0 mm

Exclusion Criteria:

* Subject is unable or is unwilling to comply with the procedural requirements of the study protocol.
* Subject has a comorbidity that in the investigator's opinion would limit life expectancy to less than 12 months.
* Subject has a known or suspected infection of the hemodialysis access site, systemic infection and/or septicemia.
* Subject has a stroke diagnosis within 3 months prior to enrollment.
* Subject has a history of unstable angina or myocardial infarction within 60 days prior to enrollment.
* Subject is pregnant, breastfeeding, or intending to become pregnant within the next year.
* Target lesion is located within a stent / stent graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects without any localized or systemic safety events (Primary Safety Endpoint | 30 days
  Proportion of subjects without any localized or systemic safety events through 30 days post-index procedure that affect the access or venous outflow circuit and resulted in intervention, hospitalization, or death.
Proportion of subjects with Target Lesion Primary Patency (TLPP) (Primary Effectiveness Endpoint) | 6 months
  Proportion of subjects with Target Lesion Primary Patency (TLPP) at 6 Months. TLPP is defined as freedom from clinically-driven target lesion revascularization (CD-TLR) or target lesion thrombosis measured through 6 months post-procedure, which is the time interval of uninterrupted patency after study procedure to the next intervention performed on the target lesion or uncorrectable target lesion occlusion.

SECONDARY OUTCOMES:
Proportion of subjects with Target Lesion Primary Patency | 12 and 24 months
Proportion of subjects with Assisted Target Lesion Primary Patency (aTLPP) | 6, 12 and 24 months
Proportion of subjects with Access Circuit Primary Patency (ACPP) | 6, 12 and 24 months
Proportion of subjects with Post-Procedure Secondary Patency | 6, 12 and 24 months
Rates of procedure- and device-related adverse events involving the access circuit | Index procedure, 30 days, and months 6, 12 and 24.

IPD SHARING:
Plan to Share IPD: No